CLINICAL TRIAL: NCT02530567
Title: Using MRI for a Non-invasive Evaluation of Portal Pressure
Brief Title: Non-invasive Evaluation of Portal Pressure by MRI
Acronym: ENIP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment defect
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RC31/14/7318; University Hospital Toulouse (Other Grant/Funding Number: 14731802)
Record Dates: First submitted 2015-08-18; First posted 2015-08-21 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Chronic Liver Disease
Keywords: portal pressure; portosystemic pressure gradient; azygos blood flow
MeSH Terms: interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental): The measurement of portosystemic pressure gradient will be performed before liver biopsy.
  Then liver biopsy is performed. The MRI was performed on the day of biopsy or within one week around the completion of the biopsy.
  The MRI machine used is the Siemens 3T.
  Interventions: Procedure: Intervention

INTERVENTIONS:
Procedure: Intervention — All patients performing the biopsy will have an MRI to carry out the necessary measures.

SUMMARY:
The objective of this research is to study the correlation between the portosystemic pressure gradient and azygos blood flow measured by MRI.

DETAILED DESCRIPTION:
All patients will benefit from:

* Pressure gradient measurement portosystemic
* MRI measurement of azygos flow, aortic, portals, spleen and lower cellar
* Liver biopsy
* Laboratory tests

ELIGIBILITY:
Inclusion Criteria:

* Suspicion of chronic liver disease
* Indication to perform a liver biopsy transjugular
* Patient able to consent

Exclusion Criteria:

* contraindication to MRI:
* Holders of a pacemaker or a defibrillator, an implanted material activated by electrical, magnetic or mechanical
* Holders of hemostatic clips intracerebral aneurysms or carotid arteries, bearing orthopedic implants
* claustrophobic
* Severe hepatic encephalopathy
* Inability to MRI in the week surrounding the first jugular

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Correlation between portosystemic pressure gradient measured by catheterization of the hepatic veins transjugular and azygos flow measured by MRI. | 1 week
  MRI and catheterization will be performed the same week.
  For the azygos blood flow (by MRI), measures will be repeated 5 times. Speed of extraction and the rate on the post processing console will be made with a double reading.
  For the measurement of portal pressure by catheterization, will be performed measurements of occluded hepatic vein pressure and free hepatic vein.
  They will be repeated 3 times each.
  These measures will be carried out to calculate the portosystemic pressure gradient.
  The flow rate and gradient measurements will be performed blindly to the other.

SECONDARY OUTCOMES:
Correlation between portosystemic pressure gradient measured by catheterization of the hepatic veins transjugular and aortic flow measured by MRI. | 1 week
  This outcome is different of primary outcome because the Measurement of azygos blood flow (MRI) is repeated on a strictly perpendicular section to the vessel facing the T4-T5 disk and the extraction speed rate and on post processing console is made by double reading.
  Measuring portal pressure by catheterization. Measurements of occluded hepatic vein pressure and free hepatic vein and will be repeated 3 times each.
  Flow measurements and gradient will be carried out blind to each other by the radiologist and the hepatologist.
Correlation between portosystemic pressure gradient measured by catheterization of the hepatic veins transjugular and throughput inferior vena measured by MRI. | 1 week
  Measurement of azygos blood flow (MRI) Repeated Measure 5 times on a strictly perpendicular cut to the vessel immediately after anastomosis of the hepatic veins to the inferior vena cava and Extraction speed and flow on post processing console with double reading.
  Measurement of portal pressure by catheterization It will be defined by the measures of occluded hepatic vein pressure and free hepatic vein and measurements will be repeated 3 times each.
  The flow rate and gradient measurements will be performed blindly to the other.

CONTACTS AND LOCATIONS:
Overall Officials: Phillipe OTAL, MD, Principal Investigator — UH TOULOUSE
Locations (1):
- UH Toulouse, Toulouse, France

REFERENCES:
- [Background] Schuppan D, Afdhal NH. Liver cirrhosis. Lancet. 2008 Mar 8;371(9615):838-51. doi: 10.1016/S0140-6736(08)60383-9. PMID 18328931
- [Background] Garcia-Pagan JC, De Gottardi A, Bosch J. Review article: the modern management of portal hypertension--primary and secondary prophylaxis of variceal bleeding in cirrhotic patients. Aliment Pharmacol Ther. 2008 Jul;28(2):178-86. doi: 10.1111/j.1365-2036.2008.03729.x. Epub 2008 May 2. PMID 18462268
- [Background] Bosch J, Abraldes JG, Berzigotti A, Garcia-Pagan JC. The clinical use of HVPG measurements in chronic liver disease. Nat Rev Gastroenterol Hepatol. 2009 Oct;6(10):573-82. doi: 10.1038/nrgastro.2009.149. Epub 2009 Sep 1. PMID 19724251
- [Background] Thabut D, Moreau R, Lebrec D. Noninvasive assessment of portal hypertension in patients with cirrhosis. Hepatology. 2011 Feb;53(2):683-94. doi: 10.1002/hep.24129. PMID 21274889